CLINICAL TRIAL: NCT04432779
Title: Impact of SARS-CoV-2 Infection During Pregnancy on Newborns and Young Children
Brief Title: Impact of COVID-19 Infection During Pregnancy on Newborns and Young Children
Acronym: ELIKYA COVID
Status: Terminated | Type: Observational
Why Stopped: Not enough financial and human resources
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Institute for Medical Immunology (IMI) (Unknown); Laboratoire Hospitalier Universitaire de Bruxelles (LHUB) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Elikya Covid
Record Dates: First submitted 2020-06-15; First posted 2020-06-16 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy; Covid-19
Keywords: Covid-19; Pregnancy; antibodies; congenital SARS infection; breast milk
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal specimens (placental tissue, serum, breast milk), Newborn specimens (umbilical cord blood)and infant specimens (serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Women tested positive to SARS-CoV-2 during pregnancy: All women who had a positive nasal swab or a positive serology during pregnancy or at delivery are included.
  Follow up end at 1 month post delivery.
  Interventions: Other: no intervention
- Women tested negative to SARS-CoV-2 during pregnancy: All women who had a positive nasal swab or a positive serology during pregnancy or at delivery are included.
  No follow up after delivery.
  Interventions: Other: no intervention
- Newborns from women tested positive: Newborns born to mothers who had a positive nasal swab or a positive serology during pregnancy or at delivery and who consented the follow up study.
  Follow up end at 3 years of age.
  Interventions: Other: no intervention
- Newborns from women tested negative: Newborns born to mothers who had no COVID-19 infection during pregnancy or at delivery and who consented the follow up study. These control children will be matched with children from the other group for gestational age and ethnicity.
  Follow up end at 3 years of age.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aim is to assess impact of COVID-19 infection during pregnancy on outcome of pregnancy, and on developement of the child in early life.

DETAILED DESCRIPTION:
All pregnant women will be tested for serology during each trimester of pregnancy and at delivery, together with a nasal swab. Children born to women with positive sawb or serology will be followed up for 3 years together with a control child born to negative mother.

In positive mothers, maternal antibodies at delivery will be characterized, placental transfer will be assessed. Persistence of antibodies in children at the age of 1 month and presence of antibodies in breast milk will be measured.

Occurence of premature birth, low birth weight, miscarriage, congenital malformations will be compared in positive and negative mothers. Follow up of children over the first 3 years of life will assess difference in susceptibility to infections and neurological developement in both groups.

ELIGIBILITY:
Inclusion Criteria:

* For pregnant women, all women who deliver in the CHU St Pierre, with oral consent.
* For children follow up: children born to positive mothers and matched controls after written consent

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women who deliver in the CHU St Pierre and children born to positive mothers and controls matched on gestational age and ethnicity
Sampling Method: Non-Probability Sample
Enrollment: 1362 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Outcome of pregnancy | Up to the delivery
  Incidence of miscarriage, premature delivery, low birth weight, preeclampsia, chorioamnionitis

SECONDARY OUTCOMES:
Prevalence of positive serology to SARS-CoV-2 at delivery | At the delivery
  Measure of antibodies in maternal serum at delivery
Transplacental transfer of antibodies to SARS-CoV-2 | At the delivery
  Measure the ratio of cord blood antibodies on maternal antibodies titers
To characterize placental alterations related to SARS-CoV-2 infection | At the delivery
  Placental histology will be performed in women tested positive for SARS-CoV-2 during pregnancy
Presence of maternal antibodies to SARS-CoV-2 in breast milk in breastfeeding mothers | At 1 month post delivery
To characterize the immunity transmitted to the newborn to cord blood and its persistence at the age of 1 month of life | Up to 1 month post delivery
  Measure of antibodies in cord blood and at the age of 1 month
Clinical evolution of the children | Up to 3 years
  Occurence of infectious disease, neurological development, growth

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Goetghebuer, MD PhD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- CHU SAINT Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dashraath P, Wong JLJ, Lim MXK, Lim LM, Li S, Biswas A, Choolani M, Mattar C, Su LL. Coronavirus disease 2019 (COVID-19) pandemic and pregnancy. Am J Obstet Gynecol. 2020 Jun;222(6):521-531. doi: 10.1016/j.ajog.2020.03.021. Epub 2020 Mar 23. PMID 32217113
- [Background] Di Mascio D, Khalil A, Saccone G, Rizzo G, Buca D, Liberati M, Vecchiet J, Nappi L, Scambia G, Berghella V, D'Antonio F. Outcome of coronavirus spectrum infections (SARS, MERS, COVID-19) during pregnancy: a systematic review and meta-analysis. Am J Obstet Gynecol MFM. 2020 May;2(2):100107. doi: 10.1016/j.ajogmf.2020.100107. Epub 2020 Mar 25. PMID 32292902
- [Background] Alzamora MC, Paredes T, Caceres D, Webb CM, Valdez LM, La Rosa M. Severe COVID-19 during Pregnancy and Possible Vertical Transmission. Am J Perinatol. 2020 Jun;37(8):861-865. doi: 10.1055/s-0040-1710050. Epub 2020 Apr 18. PMID 32305046
- [Background] Muldoon KM, Fowler KB, Pesch MH, Schleiss MR. SARS-CoV-2: Is it the newest spark in the TORCH? J Clin Virol. 2020 Jun;127:104372. doi: 10.1016/j.jcv.2020.104372. Epub 2020 Apr 14. PMID 32335336
- [Background] Dauby N, Goetghebuer T, Kollmann TR, Levy J, Marchant A. Uninfected but not unaffected: chronic maternal infections during pregnancy, fetal immunity, and susceptibility to postnatal infections. Lancet Infect Dis. 2012 Apr;12(4):330-40. doi: 10.1016/S1473-3099(11)70341-3. Epub 2012 Feb 24. PMID 22364680
- [Background] Goetghebuer T, Smolen KK, Adler C, Das J, McBride T, Smits G, Lecomte S, Haelterman E, Barlow P, Piedra PA, van der Klis F, Kollmann TR, Lauffenburger DA, Alter G, Levy J, Marchant A. Initiation of Antiretroviral Therapy Before Pregnancy Reduces the Risk of Infection-related Hospitalization in Human Immunodeficiency Virus-exposed Uninfected Infants Born in a High-income Country. Clin Infect Dis. 2019 Mar 19;68(7):1193-1203. doi: 10.1093/cid/ciy673. PMID 30215689
- [Background] McHenry MS, McAteer CI, Oyungu E, McDonald BC, Bosma CB, Mpofu PB, Deathe AR, Vreeman RC. Neurodevelopment in Young Children Born to HIV-Infected Mothers: A Meta-analysis. Pediatrics. 2018 Feb;141(2):e20172888. doi: 10.1542/peds.2017-2888. PMID 29374109
- [Background] Vohr BR, Poggi Davis E, Wanke CA, Krebs NF. Neurodevelopment: The Impact of Nutrition and Inflammation During Preconception and Pregnancy in Low-Resource Settings. Pediatrics. 2017 Apr;139(Suppl 1):S38-S49. doi: 10.1542/peds.2016-2828F. PMID 28562247
- [Background] Sutton D, Fuchs K, D'Alton M, Goffman D. Universal Screening for SARS-CoV-2 in Women Admitted for Delivery. N Engl J Med. 2020 May 28;382(22):2163-2164. doi: 10.1056/NEJMc2009316. Epub 2020 Apr 13. No abstract available. PMID 32283004